CLINICAL TRIAL: NCT04920994
Title: Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) in Comparison to Subcostal Transverse Abdominis Plane Block (TAP) in Major Abdominal Surgeries
Brief Title: Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) in Major Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Modified TAPA Block
Record Dates: First submitted 2021-06-03; First posted 2021-06-10 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Abdominal Surgery
Keywords: Thoracoabdominal nerve block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (M-TAPA ) (Active Comparator): Ultrasound-guided M-TAPA block will be performed under strict aseptic conditions with the patient in the supine position, and bupivacaine will be administered.
  Interventions: Procedure: M-TAPA block; Drug: Bupivacaine Hydrochloride
- Group B (SCTAP) (Active Comparator): Ultrasound-guided SCTAP block will be performed under strict aseptic conditions with the patient in the supine position, and bupivacaine will be administered.
  Interventions: Procedure: SCTAP block; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Procedure: M-TAPA block — A high-frequency linear ultrasound probe will be used, probe will be placed on the costochondral angle in the sagittal plane and angled deeply to view the lower aspect of the chondrium in the midline, then using in-plane approach, a 22 Gauge Tuohy needle will be introduced into the lower aspect of the chondrium. The same procedure will be repeated on the contralateral side.
  Other Names: Ultrasound guided block
  Arms: Group A (M-TAPA )
Procedure: SCTAP block — A high-frequency linear ultrasound probe will be placed obliquely on the upper abdominal wall, along the subcostal margin near the midline. After identifying the rectus abdominis muscle, the ultrasound probe will be gradually moved laterally along the subcostal margin until the transversus abdominis muscle will be identified lying posterior to the rectus muscle, then using in-plane approach, a 22 Gauge Tuohy needle will be introduced medially and directed towards the transversus abdominis plane until its tip reaches the fascia between the rectus abdominis and the transverse abdominis muscles on entering the neurofascial plane. The same procedure will be repeated on the contralateral side.
  Other Names: Ultrasound guided block
  Arms: Group B (SCTAP)
Drug: Bupivacaine Hydrochloride — 20 ml 0.25% bupivacaine will be injected after the negative aspiration test.
  Other Names: Marcaine

SUMMARY:
This study will be conducted to evaluate efficacy of ultrasound guided modified thoracoabdominal nerves block via a new perichondrial approach (M-TAPA) for postoperative analgesia in major abdominal surgeries in comparison to subcostal transverse abdominis plane (SCTAP) block.

It is hypothesized that M-TAPA block will be advantageous to SCTAP block as a promising effective alternative for analgesia for major abdominal surgeries with fewer side effects.

DETAILED DESCRIPTION:
Postoperative pain management for major abdominal surgeries can reduce postoperative respiratory dysfunction and promote early mobilization. Traditionally, opioids have been used to manage postoperative pain. However, an increasing awareness of opioid-related adverse events including respiratory depression, paralytic ileus, and sedation, has led to a shift towards utilizing opioid-sparing techniques for postoperative analgesia. As such, outcomes associated with the transverse abdominis plane block are of increasing interest. A modified thoracoabdominal nerves block via a new perichondrial approach (M-TAPA) is a novel analgesic technique that involves local anesthetic injection into the lower aspect of the chondrium. It can block thoracoabdominal nerves at T5 in cephalic direction and down to T11-T12 in caudal direction and may be an effective analgesic for major abdominal surgeries.

The aim of this study is to assess the quality of pain relief in patients who will undergo major abdominal surgery receiving either (M-TAPA) block or (SCTAP) block by comparing and evaluating the differences between the two techniques.

This prospective, randomized, comparative clinical study will include 80 patients who will be scheduled for major abdominal surgery under general anesthesia in Mansoura university hospitals. Informed written consent will be obtained from all subjects in the study after ensuring confidentiality. Eligible patients will be randomly assigned to 2 equal groups (M-TAPA group and SCTAP group) according to computer-generated table of random numbers using the permuted block randomization method. The collected data will be coded, processed, and analyzed using SPSS program. All data will be considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I and II patients.
* Scheduled for elective major abdominal surgeries.

Exclusion Criteria:

* Patient's refusal.
* Altered mental status or un-cooperative patients.
* History of known sensitivity to the used anesthetics.
* Bleeding or coagulation diathesis.
* Infection at the injection site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Total analgesic requirements of morphine | Up to 24 hours after the procedure
  The amount of morphine consumption in milligrams given as a rescue analgesia

SECONDARY OUTCOMES:
Improvement in pain scores by Visual analogue scale (VAS) | Up to 24 hours after the procedure
  VAS score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain) will be assessed postoperatively at 1, 2, 4, 8, 12, 24 hours
Duration for the first analgesic request | Up to 24 hours after the procedure
  The time of the first analgesic request for morphine in minutes will be recorded.
Changes in heart rate | Up to 24 hours after the procedure
  Heart rate (beat/min) will be recorded at baseline, intraoperative fifteen-minute intervals, 1, 2, 4, 8, 12, 24 hours postoperatively
Changes in mean arterial blood pressure | Up to 24 hours after the procedure
  Blood pressure (mmHg) will be recorded at baseline,intraoperative fifteen-minute intervals,1, 2, 4, 8, 12, 24 hours postoperatively
Incidence of adverse effects | Up to 24 hours after the procedure
  Any adverse effects like pneumothorax, respiratory depression, nausea, vomiting, pruritus, hematoma, or allergic reactions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M El-Sherbiny, MD, Principal Investigator — Mansoura Faculty of Medicine
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No